CLINICAL TRIAL: NCT02032537
Title: Efficacy of Calmmax Cream in the Management of Chronic Uremic Pruritus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Linda Shavit, Dr, Shaare Zedek Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shavit.ctil
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Calmmax Cream on UP in CKD Patients.
Keywords: callmax cream; uremic pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Callmax cream (Active Comparator)
  Interventions: Drug: Callmax cream application over affected skin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Callmax cream application over affected skin — Callmax cream application over affected skin Callmax cream or topical water containing emollient (placebo) will be applied by the patient on the affected skin area whenever the pruritus starts including night time. The frequency of application will be regulated by individual patients and increased according to pruritus severity.
  Arms: Callmax cream
Drug: Placebo — Topical water containing emollient (placebo) will be applied by the patient on the affected skin area whenever the pruritus starts including night time. The frequency of application will be regulated by individual patients and increased according to pruritus severity. The data on efficacy, duration of effect and frequency of application will be collected.during the study.
  Arms: Placebo

SUMMARY:
Uraemic pruritus (UP) remains a frequent and distressing problem in patients with advanced chronic kidney disease (CKD) and end-stage renal disease (ESRD).

Calmmax is a new topical cream that was introduced recently by Calmmax Pharma, an Israeli pharmaceutical company developed a topical cream based on active plant extracts for treatment of skin inflammation. We intend to conduct a prospective, double blind, placebo controlled, randomized trial that will assess the therapeutic effect of Calmmax cream on UP in a cohort of CKD and ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

1. History of pruritus of >8 weeks duration.
2. Severity score of pruritus ≥5 as defined by VAS
3. Discontinuation of any medication with presumed antipruritic effects at least 1 week before the study (including Calmmax cream)
4. Negative pregnancy test result for all participating women of childbearing age;

Exclusion Criteria:

1. Known allergy to Calmmax cream
2. Any acute illness
3. Liver cirrhosis
4. Active dermatological disorder other than UP
5. Decompensated heart failure
6. Inability to give informed consent
7. Known poor adherence to medical recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of UP measured by reduction of VAS by more than 50 percent from baseline score | 1 year

SECONDARY OUTCOMES:
quality of life assessed by questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Itzchak Slotki, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264